CLINICAL TRIAL: NCT04401917
Title: Evaluation of in Vivo Neuroinflammation Using 18F-NOS Positron Emission Tomography (PET/CT) in HIV Positive and Negative Subjects With Opioid Use Disorder and Healthy Controls
Brief Title: Evaluation of Neuroinflammation FNOS PET/CT in HIV (+) and (-) Subjects With OUD and Healthy Controls
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 842717
Record Dates: First submitted 2020-05-13; First posted 2020-05-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: HIV Infections; Opioid Use
MeSH Terms: conditions — HIV Infections | interventions — Fluorine-18

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- HIV positive (HIV+) subjects with Opioid Use Disorder (OUD) (Other): HIV positive (HIV+) subjects with Opioid Use Disorder (OUD): HIV+/OUD+
  Interventions: Drug: [18F]NOS
- HIV negative (HIV-) subjects with OUD (Other): HIV negative (HIV-) subjects with OUD: HIV-/OUD+
  Interventions: Drug: [18F]NOS
- HIV Positive (HIV+) subjects with OUD negative (Other): HIV+ subjects who may have been opioid-exposed but do not have current or past OUD
  Interventions: Drug: [18F]NOS
- Healthy volunteer (Other): HIV-, OUD- healthy controls who have been opioid-exposed but do not have current or past OUD
  Interventions: Drug: [18F]NOS

INTERVENTIONS:
Drug: [18F]NOS — Participants will undergo approximately 60 minutes of dynamic whole-body scanning, including the brain, starting at approximately the time of injection of [18F]NOS. PET/CT imaging sessions will include an injection of ≤ 6.5 mCi (approximate range for most studies is anticipated to be 3.5-6.5 mCi) of [18F]NOS.
  Other Names: [18F]-6-(2-fluoro-propyl)-4-methylpyridin-2-amine

SUMMARY:
The purpose of this research is to measure the extent of inflammation in the brain between different groups of participants using a radioactive tracer called [18F]NOS. A radioactive tracer is a type of imaging drug that is labeled with a radioactive tag and injected into the body. This study will see how the tracer is taken up in the brain using an imaging scan called Positron Emission Tomography / Computed Tomography (PET/CT).

Participants will undergo approximately 60 minutes of dynamic scanning of the brain starting at approximately the time of injection of [18F]NOS.

Participants are required to have a brain MRI performed within 1 year prior to study enrollment, or if the subject has not had a brain MRI that is deemed acceptable for use for this study they will be asked to undergo a research brain MRI after they have consented for this study.

DETAILED DESCRIPTION:
Opioids have direct effects on immune function and opioid receptors are expressed on immune cells, including T cells, B cells, macrophages, and microglia (3, 4). There is abundant evidence that opioids dysregulate CNS immune function (5-7). However, opioids' effects on immune function are complex, with both pro-inflammatory and immune suppressive effects having been reported (8, 9). Although the immunosuppressive effects of opioids can increase susceptibility to infection (6, 7), individuals with Opioid Use Disorder (OUD) have also been found to have higher levels of inflammation than healthy controls (HCs) (10, 11). Opioids have also been shown to enhance the expression of inducible nitric oxide synthase (iNOS), a marker of oxidative stress, effects that are reversed by NOS inhibitors and in iNOS knockout mice (12, 13). Increased expression of iNOS may also be a marker of morphine-induced microglial activation and long-term neurochemical changes in the brains of individuals with OUD may be due to elevated cytokine and NO levels via iNOS expression (14).

OUD is frequently accompanied by syndemic comorbidities, such as HIV infection (15). HIV infection itself is associated with neuroinflammation, even among patients receiving antiretroviral therapy (ART) (16-18). Thus, HIV may exacerbate the inflammatory effects of OUD (19). Indeed, morphine treatment alone decreases expression of iNOS by microglia (vs. control), but morphine and HIV in combination substantially increase iNOS expression beyond the effect of HIV alone (20). This study proposes to use [18F]NOS PET/CT imaging to evaluate neuroinflammation in HIV-positive and HIV-negative subjects with OUD, HIV-positive subjects without OUD, and HCs.

In dynamic PET/CT, kinetic analysis of the dynamic time-course of the radiotracer uptake is used to help distinguish delivery of the radiotracer from retention. For quantitation of dynamic studies, the time-course of uptake is most accurately determined when there is direct information available about the time-course of the radiotracer in the blood. This information is used to delineate the data obtained from PET imaging and can lead to better image-derived variables for study. The gold standard for kinetic modeling relies on having the time-course of the radiotracer in the arterial blood as an input to create an arterial input function (AIF) (21). To obtain direct arterial blood measurements, an arterial catheter is commonly placed in the radial artery of the wrist. Short-term arterial catheterization in healthy research subjects was reported to be safe with a low incidence of complications in 1,132 radial artery catheterizations performed for the purpose of PET research protocols (1 instance of symptomatic thrombotic occlusion was documented and resolved without intervention within weeks of the occurrence) by Everett et al (22).

Arterial catheterization is a laborious procedure requiring specialized training and often discourages people from participating in clinical studies. There may be alternative methods of creating an input function using venous blood sampling and/or image-derived input functions utilizing more limited blood sampling. Generally, arterial tracer kinetics are different from venous kinetics (23). It may be possible to substitute venous samples for arterial samples when taken during a transient equilibrium phase. Because the time at which this equilibrium is reached differs between tracers and often between species, it cannot be generalized. Thus, there is a limited time window of variable length that must be assessed individually for each new radiotracer by first sampling arterial blood to allow for correlation of the time course information. In addition, almost all radiotracers used in brain imaging produce variable amounts of radiometabolites. Imaging alone cannot distinguish the parent compound from its radioactive metabolites and plasma radioactivity from that of whole blood, and in most cases it is necessary to collect blood samples to correct for metabolites when performing kinetic modeling of image data. One potential way to estimate radiometabolite concentrations without arterial sampling is by using late venous blood samples, when the metabolite concentration is maximal and arterio-venous equilibrium has been reached. This approach must be validated for each new radiotracer as the relative concentrations of radiometabolites in venous and arterial blood may differ significantly and, therefore, venous samples do not accurately estimate arterial metabolite concentrations (21). However, whole-body dynamic imaging scans may not require arterial blood as an input to create an AIF, and consequently, venous blood can be used as an alternative to measure metabolites when the arterial blood pool is within the imaging field of view. Venous blood sampling is the preferred approach when working with some populations (e.g., IV drug users).

ELIGIBILITY:
INCLUSION CRITERIA

Cohort A (HIV+/OUD+):

1. 18-65 years of age
2. Informed of the investigational nature of this study and able to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.
3. OUD positive (+): Participants will meet DSM-5 criteria for lifetime OUD and will be on a stable dosage of OUD treatment for at least four weeks prior to the screening visit.
4. HIV positive (+): Diagnosed with HIV-1 infection per medical record review. Requirements for study participation for HIV+ participants:

   * On stable ART regimen (no changes to treatment within 4 weeks of the Screening visit)
   * Viral load of less than or equal to 200 cells/mm3 within 12 months of screening (per medical record review)
   * CD4+ count greater than 200 cells/mm3 within 12 months of screening (per medical record review)

Cohort B (HIV-/OUD+):

1. 18-65 years of age
2. Informed of the investigational nature of this study and able to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.
3. OUD positive (+): Participants will meet DSM-5 criteria for lifetime OUD and will be on a stable dosage of OUD treatment for at least four weeks prior to the screening visit.
4. HIV negative (-): Negative HIV status will be confirmed by an on-site rapid HIV test at screening.

Cohort C (HIV+/OUD-):

1. 18-65 years of age
2. Informed of the investigational nature of this study and able to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.
3. OUD negative (-): During the past year, must not meet criteria for lifetime OUD (as per DSM-5) and cannot have used an opioid for any reason in the past 30 days prior to screening as evidenced by self-report, medical record review, and urine drug testing at screening.
4. HIV positive (+): Diagnosed with HIV-1 infection per medical record review. Requirements for study participation for HIV+ participants:

   * On stable ART regimen (no changes to treatment within 4 weeks of the Screening visit)
   * Viral load of less than or equal to 200 cells/mm3 within 12 months of screening (per medical record review)
   * CD4+ count greater than 200 cells/mm3 within 12 months of screening (per medical record review)

Cohort D (HIV-/OUD-, Healthy Controls):

1. 18-65 years of age
2. Informed of the investigational nature of this study and able to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.
3. OUD negative (-): Must not meet criteria for lifetime OUD (as per DSM-5) and cannot have used an opioid for any reason in the past 30 days prior to screening as evidenced by self-report, medical record review, and urine drug testing at screening.
4. HIV negative (-): Negative HIV status will be confirmed by an on-site rapid HIV test at screening.

EXCLUSION CRITERIA

1. Women who are pregnant or breast feeding will not be eligible for this study; a urine pregnancy test will be performed in women of child-bearing potential at the screening visit and within one day of the PET/CT scan.
2. At screening, the participant's weight is > 350 lb.
3. Subjects who report claustrophobia, which in the opinion of an investigator would interfere with acquisition of the structural MRI required for PET co-registration, and/or the PET scan itself.
4. Contraindications to MRI (e.g., metal in the body that cannot be removed and is not MRI compatible). An MRI screening form will be completed during screening.
5. Screening lab values that indicate significant organ dysfunction that in the opinion of an investigator could compromise participant safety or successful participation in the study.
6. History of epilepsy or seizure disorder as assessed by medical record review and/or self-report
7. History of head trauma that in the opinion of an investigator may interfere with the uptake of applicable radiotracer as assessed by medical record review and/or self-report
8. History of schizophrenia or psychotic disorder DSM-5 diagnosis
9. Current psychiatric disorder (bipolar, schizophrenia, eating disorder and major depression with suicidal ideation, or psychotic features) identified by clinical examination or the structured interview that could interfere with study participation or make it hazardous for the subject.
10. Self-reported current alcohol consumption of greater than or equal to 15 standard drinks per week on average 30 days prior to screening visit
11. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
12. Any current medical condition, illness, or disorder as assessed by medical record review and/or self-report that is considered by a physician or investigator to be a condition that could compromise participant safety or successful participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2026-12-07 (Estimated); Study Completion 2026-12-07 (Estimated)

PRIMARY OUTCOMES:
Comparing the patterns of [18F]NOS brain uptake in OUD+ vs. OUD- subjects using PET/CT scan | 3 years
  comparing the patterns of [18F]NOS brain uptake in OUD+ vs. OUD- subjects using PET/CT scan. Comparing the whole brain [18F]NOS DVR response using a two-way ANCOVA. The primary factors in the model will be two two-level factors, one indicating presence/absence of OUD, and the other presence/absence of HIV.
Comparing the patterns of [18F]NOS brain uptake in HIV+ vs. HIV- subjects using PET/Ct scna | 3 years
  Comparing the patterns of [18F]NOS brain uptake in HIV+ vs. HIV- using PET/CT scan. Comparing the whole brain [18F]NOS DVR response using a two-way ANCOVA. The primary factors in the model will be two two-level factors, one indicating presence/absence of OUD, and the other presence/absence of HIV.
Compare patterns of [18F]NOS brain uptake as a function of the interaction of OUD and HIV status. | 3 years
  compare patterns of [18F]NOS brain uptake as a function of the interaction of OUD and HIV status

SECONDARY OUTCOMES:
Compare patterns of [18F]NOS brain uptake in regions implicated in HIV and OUD | 3 years
  The magnitude of inducement of NOS due to OUD or HIV as measured in uptake of [18F]NOS will be estimated as the absolute difference in SUV or VT values from the corresponding left and right brain regions.
Comparing peripheral blood inflammatory biomarkers as a function of both the main and interactive effects of OUD and HIV status | 3 years
  using the peripheral blood inflammatory biomarkers collected during the PET/CT scan and comparing this biomarker as a function of both the main and interactive effects of OUD and HIV status.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Dubroff, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States